CLINICAL TRIAL: NCT05106530
Title: Arrhythmogenic Risk Assessment in Coronary Artery Ectasia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mark Mohsen Nady Kamel, Resident at Cardiology Department, Assiut University
Other Study IDs: Arrhythmias in CAE patients
Record Dates: First submitted 2021-10-01; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Ectasia
Keywords: Coronary artery ectasia
MeSH Terms: conditions — Coronary Aneurysm | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary Artery Ectasia patients
  Interventions: Diagnostic Test: Holter, ECG
- Normal coronary artery patients
  Interventions: Diagnostic Test: Holter, ECG

INTERVENTIONS:
Diagnostic Test: Holter, ECG — Incidence of arrhythmias in Holter monitoring among coronary artery ectasia patients as compared to normal coronary artery patients.

SUMMARY:
The investigators thought to explore arrhythmias outcome - hidden arrhythmias, ECG features: Tp-Te interval and Tp-Te/QTc ratio, fQRS among patients with coronary artery ectasia as compared to normal coronary artery patients.

DETAILED DESCRIPTION:
All patients will be subjected to:

A. Full history taking:

- Including age, sex, history of DM, HTN, dyslipidemia and Body surface area.

B. Holter monitoring for 24 hours:

* Heart rate variability
* Hidden arrhythmias
* Hidden ischemia by monitoring ST segment changes

C. Twelve lead ECG:

* fQRS in baseline ECG
* QT dispersion.
* Tp-Te interval and Tp-Te/QTc ratio
* Tp-Te dispersion

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected CAD who are referred for elective coronary angiography and/or interventions

Exclusion Criteria:

1. Patients with a history of cardiomyopathy and myocardial infarction (MI), left ventricular hypertrophy (LVH), pathological Q wave on ECG, typical left bundle block or right bundle block, incomplete right bundle block, or paced rhythm on ECG.
2. Patients with severe renal impairment
3. Post CABG patients
4. Patients of acute coronary syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include consecutive eligible patients recruited in Assiut University Heart Hospital
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Precence of arrhythmias in 24 hours Holter monitoring | 1 year
  Incidence of arrhythmias in Holter monitoring among coronary artery ectasia patients as compared to normal coronary artery patients.

SECONDARY OUTCOMES:
• Heart rate variability in Holter monitoring | 1 year
  Heart rate variability in Holter monitoring among coronary artery ectasia patients as compared to normal coronary artery patients.
• Silent ischemia as detected by Holter | 1 years
  Presence pf ischemia in Holter monitoring among coronary artery ectasia patients as compared to normal coronary artery patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abd El Hameed, Assistant Professor, Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided